CLINICAL TRIAL: NCT06473337
Title: Vitamin D Deficiency as Independent Predictor for Plaque Vulnerability and All-cause Mortality in Patients With Symptomatic Carotid Artery Stenosis
Brief Title: Vitamin D Deficiency as Independent Predictor for Plaque Vulnerability
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stephanie Kampf, MD, Principal Investigator, Medical University of Vienna
Other Study IDs: 2449/2020
Record Dates: First submitted 2024-06-04; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Vitamin D Deficiency; Carotid Artery Diseases
MeSH Terms: conditions — Vitamin D Deficiency; Carotid Artery Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample — Serum blood sample for Vitamin D testing

SUMMARY:
Role of vitamin D in cardiovascular disease is controversial. Here the investigators aimed to investigate the association of vitamin D deficiency and carotid plaque morphology as well as outcome of participants with high-grade carotid artery stenosis undergoing carotid endarterectomy.

332 consecutive participants undergoing carotid endarterectomy for symptomatic or asymptomatic carotid artery stenosis, were prospectively included in the study, and vitamin D levels were determined prior to surgery using chemiluminescence-immunoassay.

DETAILED DESCRIPTION:
Role of vitamin D in cardiovascular disease is controversial. Here the investigators aimed to investigate the association of vitamin D deficiency and carotid plaque morphology as well as outcome of participants with high-grade carotid artery stenosis undergoing carotid endarterectomy.

332 consecutive participants undergoing carotid endarterectomy for symptomatic or asymptomatic carotid artery stenosis, were prospectively included in the study, and vitamin D levels were determined prior to surgery using chemiluminescence-immunoassay.

There is insufficient data on cardiovascular outcome in participants with CAS and vitamin D deficiency. Vitamin D would be an easily modifiable factor.

Primary goal was to investigate the influence of vitamin D levels on plaque vulnerability, major adverse cardiovascular events (MACE) and all-cause mortality in patients with carotid artery disease undergoing carotid endarterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Carotid arteriostenosis
* Patient eligible for carotid artery surgery

Exclusion Criteria:

* Oncologic disease
* Patients with hemorrhagic, lacunar or cardioembolic stroke

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carotid arteriosclerosis willing to perform surgery
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Vitamin D levels and its correlation with plaque vulnerability | through study completion, an average of 1 year
  Vitamin D levels and its correlation with plaque vulnerability is the primary outcome measurement. Serum 25-hydroxy-vitamin D is measured by the Liaison Total 25-Hydroxy-Vitamin D chemiluminescence immunoassay (CLIA) on Liaison XL immunology analyzers (DiaSorin, Saluggia, Italy.

SECONDARY OUTCOMES:
Vitamin D levels and its correlation with cardiac outcome | through study completion, an average of 1 year
  Vitamin D levels and its correlation with cardia outcome is the secondary outcome measurement. Serum 25-hydroxy-vitamin D is measured by the Liaison Total 25-Hydroxy-Vitamin D chemiluminescence immunoassay (CLIA) on Liaison XL immunology analyzers (DiaSorin, Saluggia, Italy.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Neumayer, MD,Prof., Study Director — Medical University of Vienna, Department of General Surgery, Division of Vascular Surgery
Locations (1):
- Department of General Surgery, Division of Vascular Surgery, Vienna, Austria